CLINICAL TRIAL: NCT01848535
Title: Effect of Galacto-Oligosaccharides Supplementation on Amoxicillin-treated Gut Microbiota From Healthy Adults : a Proof of Principal Study
Brief Title: Effect of GOS Supplementation on Amoxicillin-treated Gut Microbiota From Healthy Adults
Acronym: GOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABRnr42438; WUR42438 (Other: wageningen university)
Record Dates: First submitted 2013-04-16; First posted 2013-05-07 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Colonic Diseases [C06.405.469.158]
Keywords: intestinal microbiota composition; intestinal microbiota activity; gastro-intestinal complains
MeSH Terms: interventions — 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GOS addition (Placebo Comparator): All subjects will receive amoxicillin (375 mg 3x per day) for 5 days. Group 1 receives a drink with GOS (2,5 g 3x per day) simultaneously to the antibiotic for 5 days and after the antibiotic treatment for another 7 days. The intervention products should be consumed at breakfast/lunch/dinner.
  Interventions: Dietary Supplement: GOS addition; Dietary Supplement: Placebo
- placebo (maltodextrine) (Placebo Comparator): All subjects will receive amoxicillin (375 mg 3x per day) for 5 days. Group 2 receives a drink with placebo, maltodextrin(2,5 g 3x per day) simultaneously to the antibiotic for 5 days and after the antibiotic treatment for another 7 days. The intervention products should be consumed at breakfast/lunch/dinner.
  Interventions: Dietary Supplement: GOS addition; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GOS addition — GOS (2.5g 3x per day) supplemented during 12 days
  Other Names: Galacto-oligosaccharide; Vivinal GOS
Dietary Supplement: Placebo — Maltodextrine(2.5g 3x per day) supplemented during 12 days
  Other Names: maltodextrine

SUMMARY:
Prebiotics are thought to be a potential means to prevent antibiotic-associated diarrhoea because of their ability to stimulate beneficial bacteria. In-vitro results showed a promising recovery of Bifidobacteria combined with an increase of Short Chain Fatty Acids (SCFA) upon Galacto-oligosaccharides (GOS) supplementation to amoxicillin-treated microbiota. As the microbiota is nowadays considered as a key factor in human health, a further understanding of the gut microbiota functioning in-vivo is essential. This understanding of the use of specific prebiotics may possibly be beneficial in the prevention or recovery of antibiotic-disturbed microbiota. As the effects of GOS supplementation on the microbiota composition and activity from healthy adults receiving amoxicillin have never been tested in-vivo, the investigators propose the current study as a proof of principle.

Objective:

To explore whether the promising effects of GOS supplementation on the composition and activity of gut microbiota from healthy adults as found by in-vitro, can also be observed in-vivo.

Study population:

10 healthy men and women volunteers, 18 - 40 yr old

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 *
* BMI: 18.5-25 kg/m2
* Stable weight over the last 6 months
* Western diet
* Availability of information about birth by caesarean section and breast-feeding
* Regular defecation (~1day)
* Healthy as judge by the participant himself
* Having signed the informed consent form

Exclusion Criteria:

* Smoking or drug use
* Pregnant (include planning to be or gave birth in the last 6 months) or lactating woman
* Using contraceptive pill
* Gastro-intestinal diseases (e.g. irritable bowel syndrome, inflammatory bowel disease)
* Traveling to an Asian, African or south American country < 6 months before the study
* Hypersensitivity or food allergy for products used in this study (e.g. Lactose, Penicillin)
* Having hepatic disease and renal failure
* Using medication other than paracetamol, acetylsalicylic acid (aspirin), hay fever, asthma
* Not willing to have the family doctor be informed about participation to the study.
* Antibiotic use < 3 months before the study
* More than 3 antibiotic treatments in the last 2 years.
* Probiotic or prebiotic use < 1 month before the study*

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Microbiota composition | evaluation between july and september 2013
  Microbiota composition of the collected faecal sample will be investigated using a phylogenetic microarray, the Intestinal-Chip. With this microarray, more than 400 species of the intestinal microbiota can be detected.
  Bifidobacteria and Lactobacillus as beneficial bacteria as well as Enterobacteriaceae and possible other pathogens (Cells/ g faecal dry weight) will also be measured using a real-time PCR with specific primers.

SECONDARY OUTCOMES:
Microbiota activity | evaluation between july and september 2013
  The Short Chain Fatty acid (SCFA) amount produced will be measured using chromatographic approaches (Gas Chromatography, High Performance Liquid Chromatography).
  The remaining GOS will be measured with High Performance Anion Exchange Chromatography (HPAEC) or with Capillary Electrophoresis -Light Induced Fluorescence, which has a better resolution than HPAEC.

OTHER OUTCOMES:
Gastrointestinal complains | during the study (26 day) via a diary

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ladirat, MSc, Principal Investigator — Wageningen University
Locations (1):
- Laboratory of Food Chemistry, Wageningen, Netherlands

REFERENCES:
- [Background] Saulnier DM, Kolida S, Gibson GR. Microbiology of the human intestinal tract and approaches for its dietary modulation. Curr Pharm Des. 2009;15(13):1403-14. doi: 10.2174/138161209788168128. PMID 19442165